CLINICAL TRIAL: NCT02144025
Title: Prevention of Ocular Graft-Versus Host Disease With Topical Cyclosporine in Recipients of Allogeneic Hematopoietic Stem Cell Transplants Performed With a Reduced Intensity Conditioning Regimen
Brief Title: Prevention of Ocular Graft-Versus-Host Disease With Topical Cyclosporine in Recipients of Allogeneic HSCT
Acronym: HSCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dra. Olga Graciela Cantu Rodriguez, Dr., Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HU-EICHO
Record Dates: First submitted 2014-05-13; First posted 2014-05-21 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Graft-Versus-Host Disease
Keywords: Ocular Graft-Versus-Host-Disease; Topical Cyclosporine
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topical cyclosporine (Experimental): This is a single arm study of patients who have received allogeneic bone marrow transplants performed with a reduced intensity conditioning regimen. In this arm, patients who are candidates to this trial, will receive topical cyclosporine twice a day for 12 months to prevent ocular graft versus host disease.
  Interventions: Drug: Cyclosporine

INTERVENTIONS:
Drug: Cyclosporine — Use of topical cyclosporine (one drop of cyclosporine in each eye, twice a day for 12 months)
  Other Names: modusik A ofteno Brand

SUMMARY:
Ocular Graft Versus Host Disease (OGVHD) is a serious potential complication of allogeneic bone marrow transplants. The usual treatment is topical cyclosporine but when the treatment is initiated the damage to the lacrimal glands has already taken place.

The present study aims to prevent OGVHD in reduced-intensity allogeneic hematopoietic transplants by using topical cyclosporine immediately after the engraftment has been achieved

DETAILED DESCRIPTION:
The patient will start using topical cyclosporine immediately after engraftment has taken place (around day 14-18 after the cell infusion) and will continue to receive it for one year.

All >18 year old patients receiving allogeneic stem cell transplants performed with a reduced intensity conditioning regimen at our center are potential candidates for the study.

The purpose of the study is to evaluate the efficacy of topical cyclosporine in prevention of ocular versus graft disease when its use is indicated immediately after the engraftment has occured.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have written consent wishing to participate in the study
* Patients who have received an allogeneic stem cell hematopoietic transplants performed with a reduced intensity conditioning regimen
* >18 year old

Exclusion Criteria:

* <18 year old
* Patients not wishing to participate in the study or have
* Patients who have received autologous stem cell hematopoietic transplants
* Patients with history of rheumatologic diseases
* Patients with a previous diagnosis of dry eye síndrome
* Patients with previous eye surgery that disrupts corenal integrity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Ocular graft versus host disease is manifested by dry eye syndrome and disruptions in corneal integrity. The study will asses the efficacy of topical cyclosporine for preventing OGVHD manifestations | 1 year after engraftment
  The patient will start using ocular topical cyclosporine at the day of engraftment (around 14-16 days after cell infusion) and will continue to use it for one year.
  The following landmarks will be evaluated:
  1. First evaluation of a new patient with the ophtalmologist: The patient will be evaluated by a qualified ophtalmologist before the allogeneic stem cell transplant with the following tests: Corneal integrity (yes or no), Schirmer test (mm), tear break up time (seconds).
  2. Immediately after engraftment has occured (around 14-16 days after cell infusion) the patient will start using topical cyclosporine and will continue to use it for one year.
  3. There will be monthly evaluations with Schirmer test to asses tear quiality and detect dry eye syndrome.
  4. Every three months the patient will have a complete optalmologic evaluation as describe before

SECONDARY OUTCOMES:
Characteristics and clinical presentation of ocular graft versus host disease in patients receiving allogeneic bone marrow transplantation using a reduced intensity conditioning regimen | 1 year
  The secondary outcome of the study is to asses the clinical characteristics of ocular graft versus host disease in patients receiving allogeneic stem cell transplants performed with a reduced intensity conditioning regimen

OTHER OUTCOMES:
Relapse of hematologic disease prior to 12 months of ocular cyclosporine use | 12 months
  Patients who relapse after hematopoietic stem cell transplant prior to 12 months of continous ocular cyclosporine use will be evaluated for signs and symptoms of ocular GVHD and will be discarded from study because it is expected that systemic cyclosporine will also be suspended.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Cantu-Rodriguez, MD, Principal Investigator — Hospital Universitario "Dr. José Eleuterio González"
Locations (1):
- Servicio de Hematologia Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No